CLINICAL TRIAL: NCT05243641
Title: Neratinib and Capmatinib Combination (Phase Ib/II) in Metastatic Breast Cancer and Inflammatory Breast Cancer Patients With Abnormal HER-family and c-Met Pathway Activity as Measured by the CELsignia Signaling Analysis Test
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor Withdrew Support
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celcuity Inc (Industry); Novartis (Industry); Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0198; NCI-2022-01130 (Other: NCI-CTRP Clinical Trials Process Registry)
Record Dates: First submitted 2022-02-01; First posted 2022-02-17 (Actual); Results first posted 2025-05-15 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Breast Cancer; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — neratinib; capmatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1b (dose escalation) (Experimental): This portion of the study will enroll a maximum of 27 patients in the dose-finding trial including the possibility of adding up to 6 additional ER+ patients in a safety assessment of aromatic inhibitor treatment
  Interventions: Drug: Neratinib; Drug: Capmatinib
- Part 2 (dose expansion) (Experimental): This portion of the study will enroll a maximum of 29 patients
  Interventions: Drug: Neratinib; Drug: Capmatinib

INTERVENTIONS:
Drug: Neratinib — Nertatinib will be supplied as 40 mg tablets, equivalent to 48.31 mg neratinib maleate.
Drug: Capmatinib — Capmatinib will be supplied at 200 mg and 150 mg tablets

SUMMARY:
This study is to learn if the combination therapy of capmatinib and neritinib can help to control metastatic or locally advanced breast cancer. Researchers also want to find the highest tolerable dose of the combination therapy of capmatinib and neritinib that can be used in this study drug combinations. The safety of this drug combination and the CELsignia MP test methodology will also be studied.

DETAILED DESCRIPTION:
This is an open-label, phase Ib/II study of neratinib plus Capmatinib in patients with metastatic breast cancer and patients with metastatic IBC.

Phase 1b - Dose Escalation of Neratinib with Capmatinib

This phase of the study will employ the Bayesian optimal interval (BOIN) design with the 3+3 design run-in, to find the MTD. The BOIN design is implemented in a simple way similar to the traditional 3+3 design, but is more flexible and possesses superior operating characteristics that are comparable to those of the more complex model-based designs, such as the continual reassessment method (CRM). The maximum sample size for dose escalation is 18. Patients are treated in cohorts of 3, beginning with Neratinib PO dose level 1 (120 mg, Dose 1-7, 160 mg, through end of treatment, see Table 2) in combination with Capmatinib PO level 1 (400 mg, see Table 3), with a maximum of 12 patients per dose. The target toxicity rate for the maximum tolerable dose (MTD) is 25%.

Phase II

Phase II will be a prospective, open label, interventional study for patients with previously treated HER2-negative metastatic breast cancer or metastatic inflammatory breast cancer. Subjects receive Capmatinib in combination with Neratinib (including an AI for patients with ER+/HER2- breast cancer). The MTD determined during Phase 1b will be used.

This portion of the trial will be conducted to assess the overall response rate (ORR) for patients treated at the MTD. The target ORR will be 25%, with unacceptable ORR as 5%. We assess the ORR using the Bayesian optimal phase 2 (BOP2) design (Zhou, Lee and Yuan, 2017).

Up to an additional 29 evaluable subjects with measurable disease will be enrolled. An interim analysis will be performed when the number of enrolled patients reaches 15.

ELIGIBILITY:
Inclusion Criteria

1. Signed Informed Consent Form (ICF) and comply with the requirements of the study protocol
2. Age ≥ 18 years.
3. ECOG performance status 0-1
4. Confirmed diagnosis of metastatic breast cancer or inflammatory breast cancer according to international consensus criteria:

   * Onset: Rapid onset of breast erythema, edema, and/or peau d'orange, and/or warm breast, with or without an underlying breast mass
   * Duration: History of such findings no more than 6 months
   * Extent: Erythema occupying at least 1/3 of whole breast
   * Pathology: Pathologic confirmation of invasive carcinoma
5. Patients who have metastatic disease which is not amenable to curative treatment with available local and systemic therapy. Patients must have received at least 1 line or up to 6 lines of therapy in the metastatic setting with at least 2 weeks washout period before the initiation of study treatment.

   i. Unless a contraindication to therapy exists, patients with ER+ breast cancer must have received prior endocrine therapy combined with a CDK4/6 inhibitor, patients with BRCA1 or BRCA2 mutations must have received prior PARP inhibitor, and patients with PD-L1+ triple negative breast cancer must have received prior immunotherapy.

   ii. Patients with HER2-positive disease must have received at least 2 regimens of anti-HER2 therapy in metastatic setting.
6. For Phase Ib, any ER, PR, and HER2 status, For Phase 2, HER2-negative per ASCO/CAP guidelines and any ER and PR status.
7. For Phase II only, Patients with measurable disease according to the Response Evaluation Criteria in Solid Tumor (RECIST, v1.1) (local or distant) and at least one metastatic lesion amenable for biopsy (core or punch)

   NOTE:

   Measurable disease: Measurable lesions are defined as those that can be accurately measured in at least one-dimension (longest diameter to be recorded) as ≥ 20mm by chest X-ray, ≥ 10mm by computed tomography (CT) scan, ≥ 10mm with calipers by clinical exam.

   Measurable malignant lymph nodes: To be considered pathologically enlarged and measurable, a lymph node must be ≥ 15mm in short axis when assessed by CT scan.

   Non-measurable disease: All other lesions (or sites of disease), including small lesions, are considered non-measurable. Bone lesions, leptomeningeal disease, ascites, pleural/pericardial effusions, lymphangitis, cutis/pulmonitis, inflammatory breast disease, and abdominal masses [not followed by CT or magnetic resonance imaging (MRI)] are considered non-measurable.
8. Left Ventricular Ejection Fraction ≥ 50% measured by MUGA scan or Echocardiogram.
9. Abnormal HER-family and c-Met signaling activity based on CELsignia MP Test results (for phase II patients only).
10. Participants must have adequate organ function including the following laboratory values at the screening visit. Screening must occur within 28 days prior to the first dose of study drug. Screening samples for hematology and serum chemistries must be drawn within 14 days prior to the first dose of study drug:

    * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L without growth factor support
    * Platelets (PLT) ≥ 75 x 10^9/L
    * Hemoglobin (Hgb) ≥ 9 g/dL
    * Calculated creatinine clearance (using Cockcroft-Gault formula) ≥ 45 mL/min
    * Total bilirubin (TBIL) ≤ ULN (upper limit of normal) with the following exception: Patients with known Gilbert disease who have serum bilirubin level ≤ 3 x ULN may be enrolled.
    * Aspartate transaminase (AST) ≤ 3 x ULN, except for participants with liver metastasis, who may only be included if AST ≤ 5 x ULN
    * Alanine transaminase (ALT) ≤ 3 x ULN, except for participants with liver metastasis, who may only be included if ALT ≤ 5 x ULN
    * Alkaline phosphatase (ALP) ≤ 5.0 x ULN
    * Asymptomatic serum amylase ≤ grade 2. Participants with grade 1 or grade 2 serum amylase at the beginning of the study must be confirmed to have no signs and/or symptoms suggesting pancreatitis or pancreatic injury (e.g., elevated P-amylase, abnormal imaging findings of pancreas, etc.)
    * Serum lipase ≤ ULN
11. Willing and able to comply with scheduled visits, treatment plan and laboratory tests. Patients who are cognitively impaired who may not be able to comply with the oral study medication schedule are excluded.

    i) Patients with ER positive (defined at ER>/=10%)breast cancer, must start (or continue) an aromatase inhibitor of physician choice during the study duration. In addition, pre-/peri-menopausal women with ER+ breast cancer will also require ovarian suppression therapy.
12. Non-English speaking subjects are eligible as long as a translator is available at the treating site.

Exclusion Criteria:

1. Concurrent anticancer therapy within 2 weeks of initiation of study treatment; except:

   i. Endocrine therapy (SERM, aromatase inhibitor, fulvestrant, medical ovarian suppression therapy) ii. Palliative radiotherapy for bone metastases < 1 week prior to study treatment
2. Unstable and symptomatic brain metastasis (Stable disease is defined as CNS radiographic study ≥ 4 weeks from completion of radiotherapy and ≥ 2 weeks from discontinuation of corticosteroids)
3. Non-hematologic adverse events from prior anticancer therapy that have not resolved to Grade ≤ 1 (CTCAE v 5.0), except for alopecia, vitiligo, pain, constipation if these symptoms existed during screening baseline.

   i. Grade 3 or above neuropathy induced from prior treatment, that is not resolved to grade 2 or below despite best supportive care
4. Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis
5. Acute exacerbations of underlying condition within the last 12 months (requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
6. Patients with known HIV infection. Testing for HIV is not required for study screening: 1) CD4+ count<350 cells/uL; or 2) had AIDS-defining opportunistic infections < 12 months
7. Known active hepatitis B (chronic or acute) or hepatitis C infection. Testing for hepatitis is not required for study screening:

   i) Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HbsAg] test and a NEGATIVE anti-HBc [antibody to hepatitis B core antigen] antibody test). Patient is eligible if anti-HBc is POSITIVE, but should sample for HBV DNA and referral to virologist to monitor for HBV reactivation ii) Patients with positive for hepatitis C virus (HCV) antibody and have positive polymerase chain reaction (PCR) for HCV RNA.
8. Severe infections within 4 weeks prior to study treatment, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
9. Signs or symptoms of infection within 2 weeks prior to study treatment per treating physician and PI judgement.
10. Concurrent oral or IV antibiotics within 5 days prior to study treatment

    * Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are allowed and eligible so long as the antibiotic is not prohibited with the study medication (See Tables 8).
11. Major surgical procedure within 28 days prior to study treatment or anticipation of need for a major surgical procedure during the course of the study.
12. Presence or history of interstitial lung disease or interstitial pneumonitis, including clinically significant radiation pneumonitis (i.e., affecting activities of daily living or requiring therapeutic intervention).
13. Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome.
14. Clinically significant, uncontrolled heart diseases.

    * Unstable angina within 6 months prior to screening
    * Myocardial infarction within 6 months prior to screening
    * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
    * Uncontrolled hypertension defined by a Systolic Blood Pressure (SBP) ≥ 160 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 100 mm Hg, with or without antihypertensive medication. Initiation or adjustment of antihypertensive medication(s) is allowed prior to screening
    * Ventricular arrhythmias
    * Supraventricular and nodal arrhythmias not controlled with medication
    * Other cardiac arrhythmia not controlled with medication
    * QTcF (QT interval corrected by Fridericia's formula) ≥ 470 ms on the screening ECG (as mean of triplicate ECG)
15. Major surgery (e.g., intra-thoracic, intra-abdominal or intra-pelvic) within 4 weeks prior (2 weeks for resection of brain metastases) to starting study therapy or who have not recovered from side effects of such procedure.
16. Unable to swallow or absorb study drugs due to impairment of GI function or GI disease e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, or malabsorption syndrome
17. Participants receiving treatment with any enzyme-inducing anticonvulsant that cannot be discontinued at least 1 week before first dose of capmatinib, and for the duration of the study.
18. Other severe, acute, or chronic medical or psychotic conditions, substance abuse or laboratory abnormalities that in the opinion of the investigator may increase the risk associated with study participation, or that may interfere with the interpretation of study results.
19. Pregnant or nursing (lactating) women
20. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for one month after stopping treatment. Highly effective contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) total hysterectomy, or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 months prior to screening). For female subjects on the study, the vasectomized male partner should be the sole partner for that subject
    * Use of injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception. Women are considered post-menopausal and not of childbearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks before study entry. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential.
21. Sexually active males will not be eligible unless they use a condom during intercourse while taking drug and for 3 months after stopping treatment and should not father a child in this period. A condom is required for all sexually active male to prevent them from fathering a child AND to prevent delivery of study treatment via seminal fluid to partner. In addition, male participants must not donate sperm for the time period specified above.
22. Participants receiving treatment with the following medications that cannot be discontinued at least 1 week prior to the start of treatment with study therapy and for the duration of the study:

    1. strong inducers of CYP3A
    2. moderate inducer of CYP3A4
    3. strong CYP3A4 inhibitor
    4. concomitant use of a moderate CYP3A4 and P-gp dual inhibitor (verapamil).
    5. proton pump inhibitor. Neratinib may be taken at least 2 hours before or 10 hours after an H2-receptor antagonist, and 3 hours after antacids.
    6. P-gp substrates (such as digoxin, dabigatran, fexofenadine) or strong P-gp inducers (such as carbamazepine, phenytoin, rifampicin, and St. John's wort).
    7. Chronic immunosuppressive therapies including systemic corticosteroids. Steroids given for physiological replacement, as anti-emetics or inhaled as well as short course of oral/topical steroids given for allergic reactions or asthma flares are allowed.
23. No prior treatment with Capmatinib, Neratinib, or other HER2 directed tyrosine kinase inhibitor (for phase II patients only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Layman, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: August 2022~ June 2023. All recruitment was done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: 11 patients were accrued and assessed for eligibility and 10 patients were assigned to the cohort.
Groups:
- Phase Ib: Dose Level 1: Neratinib 120 mg Dose 1-7, 160 mg through end of treatment once daily + Capmatinib 400 mg twice daily
- Phase Ib: Dose Level 2: Neratinib 120 mg Dose 1-7, 160 mg Dose 8-14, 200 mg through end of treatment once daily + Capmatinib 400 mg twice daily"
- Phase Ib: Dose Level 3: Neratinib 120 mg Dose 1-7, 160 mg Dose 8-14, 240 mg through end of treatment once daily + Capmatinib 400 mg twice daily
- Phase Ib: Dose Level-1: Neratinib 120 mg Dose 1-7, 160 mg through end of treatment once daily + Capmatinib 300 mg twice daily
- Phase Ib: Dose Level-2: Neratinib 120 mg through end of treatment once daily + Capmatinib 200 mg twice daily
- Phase II: Subjects receive neratinib and capmatinib. The MTD determined during Phase Ib will be used.
Period: Overall Study
Arm/Group | Phase Ib: Dose Level 1 | Phase Ib: Dose Level 2 | Phase Ib: Dose Level 3 | Phase Ib: Dose Level-1 | Phase Ib: Dose Level-2 | Phase II
Started | 7 | 0 | 0 | 3 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 0 | 0 | 3 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0 | 1 | 0 | 0
Not completed — Disease progression | 4 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants treated. The study was terminated during phase Ib, resulting in no patient enrollment for phase II.
Groups:
- Phase Ib: Dose Level 2: Neratinib 120 mg Dose 1-7, 160 mg Dose 8-14, 200 mg through end of treatment once daily + Capmatinib 400 mg twice daily
- Total: Total of all reporting groups
Arm/Group | Phase Ib: Dose Level 1 | Phase Ib: Dose Level 2 | Phase Ib: Dose Level 3 | Phase Ib: Dose Level-1 | Phase Ib: Dose Level-2 | Phase II | Total
Number analyzed (Participants) | 7 | 0 | 0 | 3 | 0 | 0 | 10
Age, Continuous [Median (Full Range); unit: Years] | 46 [37 to 50] |  |  | 39 [34 to 62] |  |  | 44.5 [34 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 |  |  | 3 |  |  | 10
  Male | 0 |  |  | 0 |  |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  |  | 1 |  |  | 2
  Not Hispanic or Latino | 6 |  |  | 2 |  |  | 8
  Unknown or Not Reported | 0 |  |  | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0 |  |  | 0
  Asian | 0 |  |  | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0 |  |  | 0
  Black or African American | 3 |  |  | 1 |  |  | 4
  White | 4 |  |  | 1 |  |  | 5
  More than one race | 0 |  |  | 1 |  |  | 1
  Unknown or Not Reported | 0 |  |  | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 |  |  | 3 |  |  | 10

OUTCOME MEASURES:

1. Primary Outcome: To Determine Maximum Tolerated Dose for Use in the Phase II Portion of the Trial
Description: This phase of the study uses the Bayesian Optimal Interval (BOIN) design with a 3+3 run-in to identify the maximum tolerable dose (MTD). Patients are treated in cohorts of 3 with a maximum of 27 participants. Starting with Neratinib PO dose level 1 (120 mg for Dose 1-7, then 160 mg) combined with Capmatinib PO level 1 (400 mg), with up to 12 patients per dose. The target toxicity rate for the MTD is 25%.
Time Frame: Cycle1 and 2, total 56 days
Population: Baseline analysis population included all participants treated.
Measure: Number; unit: Dose level (mg)
Groups:
- Phase Ib: All participants who received Neratinib 120 mg Dose 1-7, 160 mg through end of treatment once daily + Capmatinib 300 mg twice daily or Neratinib 120 mg Dose 1-7, 160 mg through end of treatment once daily + Capmatinib 400 mg twice daily
Arm/Group | Phase Ib
Number analyzed (Participants) | 10
Dose level (mg) | NA — No MTD was determined since the study was terminated prematurely during phase Ib.

2. Primary Outcome: To Determine Overall Response Rate
Description: The overall response rate (ORR) for patients treated at the MTD in Phase II was assessed. ORR was defined as the proportion of patients who achieved a partial response or complete response as their best response. All tumor responses were evaluated according to RECIST 1.1 criteria and measured using the QIAC system.
Time Frame: Up to 3 years
Population: Patients treated at the MTD in phase II were intended to be evaluated. However, due to the study's termination during Phase Ib, no patients were analyzed for this objective.
Arm/Group | Phase II
Number analyzed (Participants) | 0

3. Secondary Outcome: To Further Characterize the Safety and Tolerability of Neratinib + Capmatinib
Description: Adverse events (AEs) graded using CTCAE version 5.0: ≥ Grade 2 for non-hematological and ≥ Grade 3 for hematological AEs observed after the first protocol intervention for phase II patients.
Time Frame: Up to 3 years
Population: as for outcome 2
Arm/Group | Phase II
Number analyzed (Participants) | 0

4. Secondary Outcome: To Determine Clinical Benefit Rate (CBR)
Description: Clinical benefit rate (CBR) is defined as the proportion of patients achieving complete response, partial response, or stable disease for ≥24 weeks, was summarized by frequency and percentage with Wilson 95% confidence intervals, overall and by dose level.
Time Frame: Up to 27 months
Population: The baseline analysis population included all treated participants. However, patients who discontinued the study due to toxicities before completing Cycle 2 and without a RECIST assessment after therapy were excluded.
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- Phase Ib: Dose Level 2: Neratinib 120 mg Dose 1-7,160 mg Dose 8-14, 200 mg through end of treatment once daily + Capmatinib 400 mg twice daily
Arm/Group | Phase Ib: Dose Level 1 | Phase Ib: Dose Level 2 | Phase Ib: Dose Level 3 | Phase Ib: Dose Level-1 | Phase Ib: Dose Level-2 | Phase II
Number analyzed (Participants) | 5 | 0 | 0 | 2 | 0 | 0
percentage | 20.0 [3.6 to 62.4] |  |  | 0.0 [0.0 to 65.8] |  |

5. Secondary Outcome: To Determine the Duration of Response (DOR)
Description: Duration of response (DOR) is defined as the period from the date of the first occurrence of a CR or PR until the first date that progressive disease or death is documented.
Time Frame: Up to 27 months
Population: Baseline analysis population included all participants treated.
Measure: Number; unit: Months
Arm/Group | Phase Ib: Dose Level 1 | Phase Ib: Dose Level 2 | Phase Ib: Dose Level 3 | Phase Ib: Dose Level-1 | Phase Ib: Dose Level-2 | Phase II
Number analyzed (Participants) | 7 | 0 | 0 | 3 | 0 | 0
Months | NA — No patient experienced partial response nor complete response, so duration of response is not estimable. |  |  | NA — No patient experienced partial response nor complete response, so duration of response is not estimable. |  |

6. Secondary Outcome: To Determine Progression Free Survival (PFS)
Description: PFS is defined as the time between date of treatment start to the date of documented disease progression or death, whichever occurs first
Time Frame: Up to 27 months
Population: Baseline analysis population included all participants treated.
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Phase Ib: Dose Level 1 | Phase Ib: Dose Level 2 | Phase Ib: Dose Level 3 | Phase Ib: Dose Level-2 | Phase II
Number analyzed (Participants) | 7 | 0 | 0 | 3 | 0
Months | 4.76 [2.13 to 7.39] |  |  | 4.54 [0.70 to 8.38] |

7. Secondary Outcome: To Determine 2 Year Overall Survival (OS)
Description: The proportion of patients in the study who are alive 2 years after enrollment on to the study
Time Frame: 2 years after enrollment
Population: All patients who received at least one dose of the study medication.
Measure: Number; unit: Percentage
Arm/Group | Phase Ib: Dose Level 1 | Phase Ib: Dose Level 2 | Phase Ib: Dose Level 3 | Phase Ib: Dose Level-1 | Phase Ib: Dose Level-2 | Phase II
Number analyzed (Participants) | 7 | 0 | 0 | 3 | 0 | 0
Percentage | 14.3 |  |  | 33.3 |  |

ADVERSE EVENTS:
Time Frame: From the initiation of the first protocol-specific intervention to 2 years following the last dose of the drug, up to 27 months.
Description: Adverse events were evaluated based on the CTCAE version 5.0. All study participants who received neratinib and capmatinib combination therapy were included in the safety analysis.
Arm/Group | Phase Ib: Dose Level 1 | Phase Ib: Dose Level 2 | Phase Ib: Dose Level 3 | Phase Ib: Dose Level-1 | Phase Ib: Dose Level-2 | Phase II
All-Cause Mortality (participants affected / at risk) | 6/7 | 0/0 | 0/0 | 2/3 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/0 | 0/0 | 1/3 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 7/7 | 0/0 | 0/0 | 3/3 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ib: Dose Level 1 (N=7) | Phase Ib: Dose Level 2 (N=0) | Phase Ib: Dose Level 3 (N=0) | Phase Ib: Dose Level-1 (N=3) | Phase Ib: Dose Level-2 (N=0) | Phase II (N=0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | NA | NA | 0 | NA | NA
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | NA | NA | 1 | NA | NA
Disease Progression (General disorders) | 0 | NA | NA | 1 | NA | NA
Lung Infection (Infections and infestations) | 0 | NA | NA | 1 | NA | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ib: Dose Level 1 (N=7) | Phase Ib: Dose Level 2 (N=0) | Phase Ib: Dose Level 3 (N=0) | Phase Ib: Dose Level-1 (N=3) | Phase Ib: Dose Level-2 (N=0) | Phase II (N=0)
Abdominal Pain (Gastrointestinal disorders) | 4 | NA | NA | 0 | NA | NA
Alanine Aminotransferase Increased (Investigations) | 3 | NA | NA | 2 | NA | NA
Alkaline Phosphatase Increased (Investigations) | 1 | NA | NA | 0 | NA | NA
Anemia (Blood and lymphatic system disorders) | 1 | NA | NA | 1 | NA | NA
Anorexia (Metabolism and nutrition disorders) | 3 | NA | NA | 1 | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | NA | NA | 1 | NA | NA
Aspartate Aminotransferase Increased (Investigations) | 2 | NA | NA | 1 | NA | NA
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | NA | NA | 0 | NA | NA
Blood Lactate Dehydrogenase Increased (Investigations) | 1 | NA | NA | 1 | NA | NA
Cardiac Disorders - Chest tightness (Cardiac disorders) | 1 | NA | NA | 1 | NA | NA
Cardiac Troponin T Increased (Investigations) | 0 | NA | NA | 1 | NA | NA
Constipation (Gastrointestinal disorders) | 3 | NA | NA | 3 | NA | NA
Creatinine Increased (Investigations) | 3 | NA | NA | 0 | NA | NA
Dehydration (Metabolism and nutrition disorders) | 4 | NA | NA | 2 | NA | NA
Diarrhea (Gastrointestinal disorders) | 6 | NA | NA | 2 | NA | NA
Dizziness (Nervous system disorders) | 3 | NA | NA | 3 | NA | NA
Ear and Labyrinth Disorders - Ear drainage (Ear and labyrinth disorders) | 1 | NA | NA | 0 | NA | NA
Edema Limbs (General disorders) | 0 | NA | NA | 1 | NA | NA
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 0 | NA | NA | 1 | NA | NA
Fall (Injury, poisoning and procedural complications) | 1 | NA | NA | 1 | NA | NA
Fatigue (General disorders) | 6 | NA | NA | 3 | NA | NA
Flu Like Symptoms (General disorders) | 1 | NA | NA | 0 | NA | NA
Headache (Nervous system disorders) | 3 | NA | NA | 1 | NA | NA
Hematuria (Renal and urinary disorders) | 2 | NA | NA | 0 | NA | NA
Hyperglycemia (Metabolism and nutrition disorders) | 1 | NA | NA | 1 | NA | NA
Hyperkalemia (Metabolism and nutrition disorders) | 0 | NA | NA | 1 | NA | NA
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | NA | NA | 0 | NA | NA
Hypocalcemia (Metabolism and nutrition disorders) | 2 | NA | NA | 1 | NA | NA
Hypoglycemia (Metabolism and nutrition disorders) | 0 | NA | NA | 1 | NA | NA
Hypokalemia (Metabolism and nutrition disorders) | 2 | NA | NA | 0 | NA | NA
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | NA | NA | 0 | NA | NA
Hyponatremia (Metabolism and nutrition disorders) | 1 | NA | NA | 2 | NA | NA
Hypotension (Vascular disorders) | 1 | NA | NA | 0 | NA | NA
Infections and Infestations - Streptococcal pharyngitis (Infections and infestations) | 0 | NA | NA | 1 | NA | NA
Insomnia (Psychiatric disorders) | 1 | NA | NA | 1 | NA | NA
Irregular Menstruation (Reproductive system and breast disorders) | 1 | NA | NA | 0 | NA | NA
Localized Edema (General disorders) | 0 | NA | NA | 1 | NA | NA
Lymphocyte Count Decreased (Investigations) | 1 | NA | NA | 1 | NA | NA
Mucositis Oral (Gastrointestinal disorders) | 1 | NA | NA | 2 | NA | NA
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 0 | NA | NA | 1 | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | NA | NA | 1 | NA | NA
Nausea (Gastrointestinal disorders) | 6 | NA | NA | 2 | NA | NA
Neutrophil Count Decreased (Investigations) | 1 | NA | NA | 1 | NA | NA
Pain (General disorders) | 1 | NA | NA | 0 | NA | NA
Paresthesia (Nervous system disorders) | 0 | NA | NA | 1 | NA | NA
Paroxysmal Atrial Tachycardia (Cardiac disorders) | 0 | NA | NA | 1 | NA | NA
Platelet Count Decreased (Investigations) | 3 | NA | NA | 1 | NA | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | NA | NA | 0 | NA | NA
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | NA | NA | 0 | NA | NA
Proteinuria (Renal and urinary disorders) | 1 | NA | NA | 1 | NA | NA
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1 | NA | NA | 0 | NA | NA
Serum Amylase Increased (Investigations) | 2 | NA | NA | 2 | NA | NA
Shingles (Infections and infestations) | 1 | NA | NA | 0 | NA | NA
Sinus Bradycardia (Cardiac disorders) | 2 | NA | NA | 0 | NA | NA
Sinusitis (Infections and infestations) | 1 | NA | NA | 0 | NA | NA
Skin and Subcutaneous Tissue Disorders - Skin lesion (Skin and subcutaneous tissue disorders) | 2 | NA | NA | 0 | NA | NA
Skin Infection (Infections and infestations) | 1 | NA | NA | 0 | NA | NA
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 | NA | NA | 0 | NA | NA
Upper Respiratory Infection (Infections and infestations) | 1 | NA | NA | 0 | NA | NA
Urinary Frequency (Renal and urinary disorders) | 1 | NA | NA | 0 | NA | NA
Urinary Tract Infection (Infections and infestations) | 2 | NA | NA | 1 | NA | NA
Urinary Urgency (Renal and urinary disorders) | 1 | NA | NA | 0 | NA | NA
Urine Discoloration (Renal and urinary disorders) | 1 | NA | NA | 0 | NA | NA
Thromboembolic event (Vascular disorders) | 0 | NA | NA | 1 | NA | NA
Vomiting (Gastrointestinal disorders) | 4 | NA | NA | 2 | NA | NA
Watering Eyes (Eye disorders) | 1 | NA | NA | 0 | NA | NA
Weight Loss (Investigations) | 2 | NA | NA | 0 | NA | NA
White Blood Cell Decreased (Investigations) | 0 | NA | NA | 1 | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/41/NCT05243641/Prot_SAP_001.pdf
  • Informed Consent Form (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/41/NCT05243641/ICF_000.pdf